CLINICAL TRIAL: NCT00298701
Title: A Randomised, Double-Blind, Placebo-Controlled, Multi-Centre Phase I Trial Investigating the Safety of GRAZAX-R in Children Aged 5-12 Years With Grass Pollen Induced Rhinoconjunctivitis (With/Without Asthma)
Brief Title: Tolerability of Grazax-R in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GT-11
Record Dates: First submitted 2006-03-01; First posted 2006-03-03 (Estimated); Last update posted 2006-05-04 (Estimated); Status verified 2006-05

CONDITIONS: Allergy
Keywords: Allergy
MeSH Terms: conditions — Hypersensitivity

INTERVENTIONS:
Biological: ALK Grass tablet

SUMMARY:
This trial is performed to assess whether the Grazax-R treatment is safe to use in children aged 5-12 years.

ELIGIBILITY:
Inclusion Criteria:

* Grass pollen induced rhinoconjunctivitis
* Boys and girls, 5-12 years of age
* Positive skin prick test to grass pollen

Exclusion Criteria:

* Previous treatment with immunotherapy

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 2006-02; Study Completion 2006-04

PRIMARY OUTCOMES:
Assessment of safety by recording of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kim Simonsen, MD, Study Director — ALK-Abelló A/S
Locations (1):
- Tangstedter Landstrasse 77, Hamburg, Germany